CLINICAL TRIAL: NCT04076670
Title: Benefits of a Psychological Intervention in Family Caregivers of Palliative Care Patients
Brief Title: A Psychological Intervention for Family Caregivers of Palliative Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, M. Antonia Pérez-Marín, Profesora Titular, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PSI2010-19426
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Palliative Care
Keywords: Intervention study; Family caregiver; Overburden; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group pf participants that received usual psychological attention.
- Experimental group (Experimental): Group of participants that received usual psychological attention plus the structured psychological intervention prosed in the study.
  Interventions: Other: Psychological intervention for family caregivers of patients at the end of life

INTERVENTIONS:
Other: Psychological intervention for family caregivers of patients at the end of life — The intervention protocol is a structured programme within the framework of counselling, that aims to reduce anxiety and depression symptoms, as well as symptoms of burden (overburden).
  Arms: Experimental group

SUMMARY:
This work aims to study the benefits a psychological intervention in family caregivers of palliative care patients can have for reducing anxiety, depression and overburden.

A parallel randomized controlled trial of two groups was performed. Information was collected on 154 family caregivers of patients at the end of life during the moments before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* To be the main family caregiver of a patient at the end of life, receiven palliative care. In the present study, the main family caregiver is defined as follows: family member who assumes the main tasks of care and attends to the patient most of the time, or for a longer period of time than other members of the family.
* To have signed the informed consent.

Exclusion Criteria:

• To present cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in anxiety (PRE and POST measures) | Baseline up to 3 months
  This variable was assesed with the Hospital Anxiety and Depression Scale, HADS. This Scale contains 7 items asessing anxiety, where lower values represent a better outcome.
  In order to observe the change in anxiety, it was measured at two time points:
  First measurement: PRE. Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: POST. Up to 3 months after the first measurement the second measurement of the same variable was carried out.
  Between first and second measurement, the control group received the usual psychological attention, whereas the intervention group received the usual psychological attention plus the structured psychological intervention proposed in this study.
Change in depression (PRE and POST measures) | Baseline up to 3 months
  This variable was assesed with the Hospital Anxiety and Depression Scale, HADS.
  In order to observe the change in depression, it was measured at two time points:
  First measurement: PRE. Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: POST. Up to 3 months after the first measurement the second measurement of the same variable was carried out.
  Between first and second measurement, the control group received the usual psychological attention, whereas the intervention group received the usual psychological attention plus the structured psychological intervention proposed in this study.
Change in burden (PRE and POST measures) | Baseline up to 3 months
  This variable was assesed with the Zarit Burden Inventory.
  In order to observe the change in burden, it was measured at two time points:
  First measurement: PRE. Once the participant had signed the informed consent, the initial score for this outcome was assessed.
  Second measurement: POST. Up to 3 months after the first measurement the second measurement of the same variable was carried out.
  Between first and second measurement, the control group received the usual psychological attention, whereas the intervention group received the usual psychological attention plus the structured psychological intervention proposed in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Barreto Martin, PhD, Principal Investigator — Universitat de València
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No